CLINICAL TRIAL: NCT02556190
Title: Colistin Pharmacokinetics in Critically Ill Patients With Acute Kidney Injury AKIN III During Extended Dialysis Using the GENIUS Dialysis System
Brief Title: Colistin Pharmacokinetics in Critically Ill Patients During Extended Dialysis
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: COL-6446-2013
Record Dates: First submitted 2015-08-24; First posted 2015-09-22 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Infection Due to Resistant Bacteria; Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * blood samples
  * dialysate samples
Oversight: Data Monitoring Committee: No

SUMMARY:
The emergence of multidrug-resistant bacteria has recently renewed interest in colistin. Data on dosing in critically ill patients undergoing extended dialysis are missing. The aim of this study is to determine the pharmacokinetics of colistin during extended dialysis in critically ill patients and to provide dosing guidelines for this drug.

DETAILED DESCRIPTION:
Due to the lack of new antibiotics for the treatment of critically ill patients with multidrug-resistant bacteria, interest in "old" antibiotics like colistin re-emerged. Lastly, colistin is administered more frequently especially in cases of infections due to Pseudomonas aeruginosa, Klebsiella pneumoniae or Acinetobacter baumanii in intensive care units (ICUs) around the world. However, dosing of colistin in critically ill patients undergoing renal replacement therapy is based on scarce data. The aim of this study is to evaluate single and multiple-dose pharmacokinetics of both colistin and its inactive prodrug colistin-methanesulfonate (CMS) in critically ill patients with acute kidney injury (AKI) undergoing extended daily dialysis (EDD).

The investigators perform a prospective clinical pharmacokinetic single- and multiple-dose study in the medical and surgical ICUs of the Hannover Medical School. ICU patients with anuric AKI being treated with EDD and receiving i.v. colistin are studied on day 1 and (if possible) on day 5-9 of treatment. A loading dose of 6 Mio IU colistin ís administered 8 hours prior to the EDD session followed by 3 Mio IU every 8 hours. Colistin Plasma concentration levels as well as dialyzer clearance rates are measured at different time points.

ELIGIBILITY:
Inclusion Criteria:

* Indication for colistin therapy
* Acute kidney injury AKIN III with need for renal replacement therapy

Exclusion Criteria:

* participation in other studies
* pregnancy
* known colistin allergy or other contraindications for colistin therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients in a tertiary hospital with acute kidney injury AKIN III with need for renal replacement and colistin therapy.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Colistin elimination during extended dialysis | Participants will be followed for 10 days. Colistin elimination measured by the total drug amount in the collected spent dialysate
  Colistin elimination during extended dialysis is measured on day 1 and day 9 after colistin therapy was started. Colistin elimination is measured by the total eliminated drug amount in the total spent dialysate

SECONDARY OUTCOMES:
Colistin peak concentration during extended daily dialysis C(max) | Participants will be followed for 10 days. Colistin concentration is measured at different time points after drug infusion: 0, 0.5, 1, 1.5, 2, 4, 6, 8) on day 1 and day 9 after therapy initiation
Colistin trough Level during extended daily dialysis C(max) | Participants will be followed for 10 days. Colistin concentration is measured at different time points after drug infusion: 0, 0.5, 1, 1.5, 2, 4, 6, 8) on day 1 and day 9 after therapy initiation
Colistin dialyzer clearance during extended dialysis | Participants will be followed for 10 days. Dialyzer clearance is calculated after 30 and 180 minutes of extended dialysis on day 1 and day 9 after therapy initiation

CONTACTS AND LOCATIONS:
Overall Officials: Jan T Kielstein, Prof, Principal Investigator — Hannover Medical School, Dep. of Nephrology and Hypertension
Locations (1):
- Hannover Medical School, Hanover, Lower Saxony, Germany

REFERENCES:
- [Derived] Schmidt JJ, Strunk AK, David S, Bode-Boger SM, Martens-Lobenhoffer J, Knitsch W, Scherneck S, Welte T, Kielstein JT. Single- and multiple-dose pharmacokinetics and total removal of colistin in critically ill patients with acute kidney injury undergoing prolonged intermittent renal replacement therapy. J Antimicrob Chemother. 2019 Apr 1;74(4):997-1002. doi: 10.1093/jac/dky511. PMID 30624668